CLINICAL TRIAL: NCT04600726
Title: Application of VR-based Working Memory Screening Test to Facilitate Early Detection of Dementia
Brief Title: Application of VR-based Working Memory Screening Test
Acronym: VR
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: The Hong Kong Polytechnic University (Other)
Collaborators: Department of Neuroscience, Psychology and Behavior. The University of Leicester (Unknown); School of Psychology, The University of Nottingham (Unknown); The Alice Ho Miu Ning Nethersole Hospital (Unknown)
Responsible Party: Principal Investigator, Dr Frank LAI, Assistant Professor, The Hong Kong Polytechnic University
Other Study IDs: VR_Clinical Trial
Record Dates: First submitted 2020-10-19; First posted 2020-10-23 (Actual); Last update posted 2020-10-23 (Actual); Status verified 2020-10

CONDITIONS: Older Adults With Mild Neurocognitive Disorders; Older Adults With Non-communicable Diseases; Healthy Age-matched Older Adults
Keywords: Cognitive function screening

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Biospecimen Retention: Samples Without DNA — The panel of biomarkers covers five immune cytokines and two metabolic markers (including serum IL-1B,Interleukin 6, Interleukin 10, Interleukin 33, Tumor Necrosis Factor alpha, Leptin and Glycosylated haemoglobin A1c (HbA1c)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- older adults with known mild NCD: Older adults with known mild neuro-cognitive disorders
  Interventions: Other: no intervention
- older adults with non-communicable diseases: older adults with non-communicable diseases such as diabetics, hypertension and chronic obstructive airway diseases
  Interventions: Other: no intervention
- Older adults with healthy condition: Older adults who are free from neuro-cognitive disorders and non-communicable diseases
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention — no interventioni

SUMMARY:
We propose to validate an interactive, immersive spatial memory test from the laboratory test. This VR-based working memory test (VRWMT) is a first-person, self-pacing game embedded within a virtual reality environment, the program is easily implemented with minimal instructions and no supervision that can be community-users friendly. It is specifically designed to assess rapid spatial working memory - a common deficit in all NCD subtypes. Its ability to detect pathological models of dementia, age-related deterioration, and hippocampal dysfunction are well established in literature

DETAILED DESCRIPTION:
The proposed research aims to study the ability of VRWMT to discriminate between older adults with known mild NCD, healthy age-matched older adults and participants with non-communicable diseases and to predict their deterioration in cognitive function over a period of 12 months. Moreover, this study is to characterize and evaluate any concurrent validity between emergence of deterioration in the VRWMT and clinical tools of functional performance in older adults. Additionally, the potential of inflammatory and metabolic dysregulation biomarkers to increase our ability to detect early NCD risk over and above the predictive validity of the VRWMT. The study findings will bring both social and clinical significance to ageing and NCD research. The combination of behavioural and biomarkers of pathological significance offers an innovative approach that potentially addresses the limitations intrinsic to either measure alone.

ELIGIBILITY:
Inclusion Criteria:

* the ability to understand verbal and written Chinese instructions
* the ability and willingness to provide informed consent and sign the relevant document.

Exclusion Criteria:

* a history of substance abuse including alcohol, drugs, or any medication/substances indicative of chronic abuse;
* participants with major NCD.

Ages: 65 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: Older adults who are community dwelling
Sampling Method: Probability Sample
Enrollment: 160 (Estimated)
Dates: Start 2021-02-01 (Estimated); Primary Completion 2022-12-30 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Delayed matching-to-place (DMP) | 20 mins
  a prototypical working memory test implemented in a virtual reality environment of the VRWMT
The Montreal Cognitive Assessment - Hong Kong Version | 15 mins
  The MoCA-HK is an examiner-rated cognitive screening test that evaluates visuospatial functions, naming, attention and working memory, language, abstraction, and orientation, commonly affected in NCD including Alzheimer's disease, stroke, and vascular dementia. It is a validated tool for detecting cognitive impairment in Chinese Hong Kong population at early stages. It is a common tool in practical practice that can be under 15 minutes. MoCA scores range from 0 to 30. Subjects with a score of above 21 will be classified as "healthy controls", while 21 or below will be included in the mild NCD group in the present study.
The Chinese Multiple Errands Test | 20 mins
  A functional performance measure of executive function that identifies abnormalities known for its ecological validity through assessment of real-world daily living activities. The proposed study will evaluate the ability of working memory (as a component to executive function) from VRWMT to predict executive functions (globally) across the six scores obtained from the Chinese Multiple Errands Test
Biological biomarkers for older adults with NCDs and Healthy Control | 5 mins
  The panel of biomarkers covers five immune cytokines and two metabolic markers (including serum IL-1B,Interleukin 6, Interleukin 10, Interleukin 33, Tumor Necrosis Factor alpha, Leptin and Glycosylated haemoglobin A1c (HbA1c)

IPD SHARING:
Plan to Share IPD: No
The data that support the findings of this study are available from the corresponding author upon reasonable request.

REFERENCES:
- [Background] Daugherty AM, Raz N. A virtual water maze revisited: Two-year changes in navigation performance and their neural correlates in healthy adults. Neuroimage. 2017 Feb 1;146:492-506. doi: 10.1016/j.neuroimage.2016.09.044. Epub 2016 Sep 19. PMID 27659539
- [Background] Daugherty AM, Bender AR, Yuan P, Raz N. Changes in Search Path Complexity and Length During Learning of a Virtual Water Maze: Age Differences and Differential Associations with Hippocampal Subfield Volumes. Cereb Cortex. 2016 Jun;26(6):2391-401. doi: 10.1093/cercor/bhv061. Epub 2015 Apr 1. PMID 25838036
- [Background] Folley BS, Astur R, Jagannathan K, Calhoun VD, Pearlson GD. Anomalous neural circuit function in schizophrenia during a virtual Morris water task. Neuroimage. 2010 Feb 15;49(4):3373-84. doi: 10.1016/j.neuroimage.2009.11.034. Epub 2009 Dec 4. PMID 19948225
- [Result] Daugherty AM, Yuan P, Dahle CL, Bender AR, Yang Y, Raz N. Path Complexity in Virtual Water Maze Navigation: Differential Associations with Age, Sex, and Regional Brain Volume. Cereb Cortex. 2015 Sep;25(9):3122-31. doi: 10.1093/cercor/bhu107. Epub 2014 May 23. PMID 24860019